CLINICAL TRIAL: NCT06416475
Title: The Effect of Wolffia Globosa (Mankai) on Glycemic Control Among Patients With Type 2 Diabetes; A 3-month Randomized Controlled Pilot Trial
Brief Title: The Effect of Mankai on Glycemic Control Among Patients With T2D
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ben-Gurion University of the Negev (Other)
Collaborators: Soroka University Medical Center (Other)
Responsible Party: Principal Investigator, Iris Shai, Prof. Iris Shai, Ben-Gurion University of the Negev
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SOR-0259-23
Record Dates: First submitted 2024-03-21; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: clinical trial; Diabetes Mellitus, Type 2; nutritional intervention; Mankai Duckweed; Wolffia-globosa; polyphenols
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Drinking

STUDY DESIGN:
Intervention Model Description: A 3-month Randomized Controlled pilot Trial among 104 patients with T2D, who will be randomly allocated to consume comparable bottle volumes of either crude plant Mankai beverage (60ml Mankai) or water (60ml) on top of a standardized MediterraneanT2D-recommended healthy diet, after morning, lunch, and dinner over 3 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mankai supplementation group (Active Comparator): Three times a day supplementation of postprandial Mankai duckweed drink (60mL crude plant Mankai beverage) right after breakfast, lunch, and dinner while maintaining the recommended Mediterranean diet lifestyle and medical treatment.
  Interventions: Dietary Supplement: Mankai supplementation
- Water group (Placebo Comparator): Three times a day consumption of postprandial water (60mL) right after breakfast, lunch, and dinner while maintaining the recommended Mediterranean diet lifestyle and medical treatment.
  Interventions: Other: Water consumption

INTERVENTIONS:
Dietary Supplement: Mankai supplementation — The overall dose of the three Mankai duckweed beverages/day contains ~10 grams of dry matter.
  Arms: Mankai supplementation group
Other: Water consumption — Water consumption
  Arms: Water group

SUMMARY:
The investigators aim to explore the effect of daily supplementation of Wolfia globosa Mankai on HbA1c and insulin resistance response among participants with type 2 diabetes (T2D). The investigators hypothesize that adding daily Mankai to T2D's healthy nutrition might lower HbA1c and promote glycemic control.

Methods: A 3-month pilot RCT among 104 patients with T2D, with two intervention arms consuming comparable bottle volumes of either crude plant Mankai beverage (60ml Mankai) or water (60ml) 3 times/day postprandially over 3 months. Blood, urine, fecal, and clinical measures will be taken at 0 and 3 months. Overall appetite, food intake, symptoms, and medical treatment will be monitored.

Importance: This study's results will shed light on the effects of regular Mankai consumption on HbA1c among patients with T2D, which may reveal a new nutritional source to improve glycemic control in T2D.

DETAILED DESCRIPTION:
Type 2 diabetes (T2D), most commonly stemming from sustained obesity, adiposity, and a sedentary lifestyle, is strongly associated with increased cardiovascular risk. Glycated hemoglobin A1c (HbA1c), reflecting glycemic control, is tightly related to cardiovascular risk. In the recent decade, several antihyperglycemic medications have been shown to modify cardiovascular risk among patients with established cardiovascular disease. Maintaining a healthy diet, preferably a Mediterranean-like diet, rich in plant-based protein and low in meat products, is the first-line intervention to promote glycemic control and reduce cardiovascular risk among T2D. However, whether specific nutritional products may independently promote glycemic control beyond medical treatment is unclear.

Mankai, a newly cultivated duckweed Wolffia-globosa strain, has been extensively studied in recent years. Mankai is rich in whole bioavailable protein, iron, and vitamin B12 and is rich in 200 different potent polyphenols, potentially affecting the metabolomic-gut-clinical axis. Mankai consumption, as a dominant part of the green-Mediterranean diet, was shown to promote weight loss, systemic inflammation lowering, and cardiometabolic risk reduction and was associated with regressions in hepatosteatosis, visceral abdominal adiposity, and proximal aortic stiffness among patients with abdominal obesity with or without T2D. Also, Mankai consumption was mainly linked with improved glycemic control, dramatic elevation in fasting Ghrelin levels, and insulin sensitivity recovery. Regular Mankai consumption promoted microbiome optimization, mainly impacting bacterial glucose metabolism and human glucose control.

In this proposed study, The investigators aim to explore the effect of daily consumption of 60mL crude plant Mankai beverage boost after 3 meals among patients with T2D on HbA1c levels (gold-standard for assessing glycemic control, primary outcome).

"Mankai" is a cultivated strain of Wolffia globosa, an aquatic plant, part of the family of plants known commonly as duckweeds. Duckweeds are elementary flowering aquatic plants floating on or beneath still or slow-moving water bodies.

There is a long history of using Wolffia species, particularly Wolffia globosa, as food, especially in Southeast Asia: Burma, Laos, and northern Thailand, where it has been used as a vegetable for many generations. The plant is cultivated locally in rain-fed open ponds, grown commercially in Thailand, and sold in local markets throughout Thailand and Laos. There are numerous ways of Wolffia globosa consumption and a variety of recipes, using it either as the main ingredient (such as Wolffia crisps or "Kaeng pum" - a popular vegetable dish in northeastern Thailand) or incorporating it in other foods (e.g., Wolffia-meat ball, fermented Wolffia-meat sausage, Wolffia rice noodle, Wolffia cookies, Wolffia bread, and various soups and salads). Moreover, Wolffia is known as one of the essential food sources in northern Thailand.

Along with its long history as a food source in Southeast Asia, it is recognized as an edible vegetable for humans in several databases, including the USDA (2014) GRIN database and a database dedicated to tropical species. For the proposed clinical trial, Mankai will be provided as a beverage, refrigerated at ±4°C. Participants will consume Mankai as an additional additive to a standardized healthy Mediterranean diet.

ELIGIBILITY:
Inclusion Criteria:

* Age > 30 years
* A formal diagnosis of T2D (126mg/dl fasting glucose or higher, or HbA1c>6.5%) or taking T2D medications with HbA1c levels over 7%
* Medication stability for at least 3 months prior to Intervention initiation
* Adherence to medical follow-up in primary care clinic or diabetes-centered outpatient services

Exclusion Criteria:

* HbA1c lower than 7% or higher than 10%
* Known insulinopenia
* Treatment with coumadin (warfarin)
* Advanced renal failure
* Significantly disturbed liver enzymes (liver transaminases or bilirubin levels more than time three upper-normal-limit)
* A significant illness that might require hospitalization
* Regular Mankai consumption
* State of pregnancy or lactation
* Presence of active cancer or chemotherapy treatment in last three years
* Participation in another trial

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2024-04-30 (Actual); Primary Completion 2024-08-08 (Estimated); Study Completion 2024-08-15 (Estimated)

PRIMARY OUTCOMES:
HbA1c | Baseline and three months time points
  Glycated hemoglobin-HbA1c; as detected by a standard laboratory measure
Fasting glycemic and insulin resistance profiling | Baseline and three months time points
  Fasting glycemic and insulin resistance profiling [using calculated homeostatic model assessment of insulin resistance (HOMA-IR) as detected by laboratory assessment]

SECONDARY OUTCOMES:
Lipid profile | Baseline and three months time points
  Changes in lipid biomarkers (blood draw), such as LDL (mg/dL), HDL (mg/dL), TG (mg/dL), total cholesterol (mg/dL), Lipoprotein (a) (mg/dL)
Lipid profile | Baseline and three months time points
  Changes in lipid biomarkers (blood draw), such as apo(A)1(g/L), apo(B)100 (g/L)
Hormones and adipokines | Baseline and three months time points
  Changes in hormone and adipokine biomarkers (blood draw); such as total adiponectin (ug/ml), RBP4 (ug/ml), chemerin (ng/ml), vaspin (ng/ml), omentin-1(ng/ml), MCP-1 (pg/ml)
Inflammatory biomarkers | Baseline and three months time points
  Changes in inflammatory biomarkers (blood draw); such as CRP (mg/dl), IL-1 (pg/mL), IL-6 (pg/mL), IL10 (pg/mL), IL-17 (pg/mL), TNF-alpha (pg/mL)
Hunger/satiety hormones | Baseline and three months time points
  Changes in Hunger/satiety hormones (blood draw); such as leptin(ng/ml), ghrelin(pg/ml), neuropeptide Y (NPY) (pg/ml), cholecystokinin (CCK) (pmol/L), peptide YY (PYY) (pmol/L), and incretins (e.g., oxyntomodulin (pmol/L) and glucagon-like peptide-1 (GLP-1)(pmol/L)]
CVD biomarkers | Baseline and three months time points
  Changes in CVD biomarkers (blood draw); such as Homocysteine (ug/dL)
CVD biomarkers | Baseline and three months time points
  Changes in CVD biomarkers (blood draw); such as Renin (iU/ml)
CVD biomarkers | Baseline and three months time points
  Changes in CVD biomarkers (blood draw); such as Troponin (cardiac troponin I and T) (ng/ml)
CVD biomarkers | Baseline and three months time points
  Changes in CVD biomarkers (blood draw); such as NT-pro-BNP (pg/ml)
Cardiometabolic health-Liver function (blood biomarkers) | Baseline and three months time points
  Changes in liver function biomarkers (blood draw); such as Alkaline Phosphatase (U/L), Alanine Aminotransferase (U/L), Aspartate Aminotransferase (U/L), bilirubin (mg/dL)
Cardiometabolic health-Liver function (blood biomarkers) | Baseline and three months time points
  Changes in liver function biomarkers (blood draw); such as bilirubin (mg/dL)
HPA axis biomarkers | Baseline and three months time points
  Changes in HPA axis biomarkers (blood draw); such as ACTH (pmol/L)
HPA axis biomarkers | Baseline and three months time points
  Changes in HPA axis biomarkers (blood draw); such as cortisol (nmol/L)
HPA axis biomarkers | Baseline and three months time points
  Changes in HPA axis biomarkers (blood draw); such as cortisone (microg/L)
HPG axis biomarkers | Baseline and three months time points
  Changes in HPG axis; such as Testosterone (nmol/L), SHBG (nmol/L), IGF1 (nmol/L)
HPG axis biomarkers | Baseline and three months time points
  Changes in HPG axis; such as LH (IU/mL)
HPG axis biomarkers | Baseline and three months time points
  Changes in HPG axis; such as FSH (IU/L)
HPG axis biomarkers | Baseline and three months time points
  Changes in HPG axis; such as GH (pmol/L)
Well being | Baseline and three months time points
  Assessed by questionnaires; 1. Screening questionnaire 2. I-MEDAS (Mediterranean Diet Adherence Screener) questionnaire - the 14-item MEDAS questionnaire (scale 0-17, higher score indicated higher adherence to Mediterranean diets), 3. Validated physical activity questionnaire, 4. Symptoms questionnaire, 5. Medical questionnaire, and 6. A follow-up questionnaire.
Microbiota profiling | Baseline and three months time points
  Shannon Diversity Index (where 0 indicates no diversity, there is no upper limit to the index, usually between 1.5 - 3.5).
Weight | Baseline and three months time points
  Bodyweight will be measured without shoes to the nearest 0.1 kg.
Waist circumference | Baseline and three months time points
  WC will be measured halfway between the last rib and the iliac crest to the nearest millimeter by standard procedures using a 150-cm anthropometric measuring tape.
BMI | Baseline and three months time points
  Weight and Height will be combined to report BMI in kg/m^2
Blood pressure | Baseline and three months time points
  Blood pressure will be measured and determined using an automated system in mmHg. Both systolic and diastolic blood pressure will be measured.
Resting pulse | Baseline and three months time points
  Pulse will be measured and determined using an automated system in Beats per minute.
Urine biomarkers | Baseline and three months time points
  Urine albumin (mg/dL)
Urine biomarkers | Baseline and three months time points
  UACR (mg/g)
Urine biomarkers | Baseline and three months time points
  Urine creatinine (g/dL)
Urine biomarkers | Baseline and three months time points
  eGFR (ml/min/1.73m^2)
Urine biomarkers | Baseline and three months time points
  Urine polyphenols for adherence as measured by mass spectrometry.

CONTACTS AND LOCATIONS:
Overall Officials: Idit Liberty, Principal Investigator — Soroka University Medical Center; Iris Shai, Study Director — Ben-Gurion University of the Negev
Locations (1):
- Soroka Medical Center, Beersheba, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Piche ME, Tchernof A, Despres JP. Obesity Phenotypes, Diabetes, and Cardiovascular Diseases. Circ Res. 2020 May 22;126(11):1477-1500. doi: 10.1161/CIRCRESAHA.120.316101. Epub 2020 May 21. PMID 32437302
- [Background] Joseph JJ, Deedwania P, Acharya T, Aguilar D, Bhatt DL, Chyun DA, Di Palo KE, Golden SH, Sperling LS; American Heart Association Diabetes Committee of the Council on Lifestyle and Cardiometabolic Health; Council on Arteriosclerosis, Thrombosis and Vascular Biology; Council on Clinical Cardiology; and Council on Hypertension. Comprehensive Management of Cardiovascular Risk Factors for Adults With Type 2 Diabetes: A Scientific Statement From the American Heart Association. Circulation. 2022 Mar;145(9):e722-e759. doi: 10.1161/CIR.0000000000001040. Epub 2022 Jan 10. PMID 35000404
- [Background] Zhu J, Yu X, Zheng Y, Li J, Wang Y, Lin Y, He Z, Zhao W, Chen C, Qiu K, Wu J. Association of glucose-lowering medications with cardiovascular outcomes: an umbrella review and evidence map. Lancet Diabetes Endocrinol. 2020 Mar;8(3):192-205. doi: 10.1016/S2213-8587(19)30422-X. Epub 2020 Jan 29. PMID 32006518
- [Background] Yancy WS Jr, Dunbar SA, Boucher JL, Cypress M, Evert AB, Franz MJ, Mayer-Davis EJ, Neumiller JJ, Urbanski P, Verdi CL, Nwankwo R. Response to comments on Evert et al. Nutrition therapy recommendations for the management of adults with diabetes. Diabetes care 2013;36:3821-3842. Diabetes Care. 2014 May;37(5):e102-3. doi: 10.2337/dc14-0077. No abstract available. PMID 24757235
- [Background] Corrigendum to: 2021 ESC Guidelines on cardiovascular disease prevention in clinical practice: Developed by the Task Force for cardiovascular disease prevention in clinical practice with representatives of the European Society of Cardiology and 12 medical societies With the special contribution of the European Association of Preventive Cardiology (EAPC). Eur Heart J. 2022 Nov 7;43(42):4468. doi: 10.1093/eurheartj/ehac458. No abstract available. PMID 36083202
- [Background] Kaplan A, Zelicha H, Tsaban G, Yaskolka Meir A, Rinott E, Kovsan J, Novack L, Thiery J, Ceglarek U, Burkhardt R, Willenberg A, Tirosh A, Cabantchik I, Stampfer MJ, Shai I. Protein bioavailability of Wolffia globosa duckweed, a novel aquatic plant - A randomized controlled trial. Clin Nutr. 2019 Dec;38(6):2576-2582. doi: 10.1016/j.clnu.2018.12.009. Epub 2018 Dec 11. PMID 30591380
- [Background] Yaskolka Meir A, Tsaban G, Zelicha H, Rinott E, Kaplan A, Youngster I, Rudich A, Shelef I, Tirosh A, Brikner D, Pupkin E, Sarusi B, Bluher M, Stumvoll M, Thiery J, Ceglarek U, Stampfer MJ, Shai I. A Green-Mediterranean Diet, Supplemented with Mankai Duckweed, Preserves Iron-Homeostasis in Humans and Is Efficient in Reversal of Anemia in Rats. J Nutr. 2019 Jun 1;149(6):1004-1011. doi: 10.1093/jn/nxy321. PMID 30915471
- [Background] Sela I, Yaskolka Meir A, Brandis A, Krajmalnik-Brown R, Zeibich L, Chang D, Dirks B, Tsaban G, Kaplan A, Rinott E, Zelicha H, Arinos S, Ceglarek U, Isermann B, Lapidot M, Green R, Shai I. Wolffia globosa-Mankai Plant-Based Protein Contains Bioactive Vitamin B12 and Is Well Absorbed in Humans. Nutrients. 2020 Oct 8;12(10):3067. doi: 10.3390/nu12103067. PMID 33049929
- [Background] Yaskolka Meir A, Tuohy K, von Bergen M, Krajmalnik-Brown R, Heinig U, Zelicha H, Tsaban G, Rinott E, Kaplan A, Aharoni A, Zeibich L, Chang D, Dirks B, Diotallevi C, Arapitsas P, Vrhovsek U, Ceglarek U, Haange SB, Rolle-Kampczyk U, Engelmann B, Lapidot M, Colt M, Sun Q, Shai I. The Metabolomic-Gut-Clinical Axis of Mankai Plant-Derived Dietary Polyphenols. Nutrients. 2021 May 30;13(6):1866. doi: 10.3390/nu13061866. PMID 34070816
- [Background] Tsaban G, Yaskolka Meir A, Rinott E, Zelicha H, Kaplan A, Shalev A, Katz A, Rudich A, Tirosh A, Shelef I, Youngster I, Lebovitz S, Israeli N, Shabat M, Brikner D, Pupkin E, Stumvoll M, Thiery J, Ceglarek U, Heiker JT, Korner A, Landgraf K, von Bergen M, Bluher M, Stampfer MJ, Shai I. The effect of green Mediterranean diet on cardiometabolic risk; a randomised controlled trial. Heart. 2021 Jun 11;107(13):1054-1061. doi: 10.1136/heartjnl-2020-317802. PMID 33234670
- [Background] Yaskolka Meir A, Rinott E, Tsaban G, Zelicha H, Kaplan A, Rosen P, Shelef I, Youngster I, Shalev A, Bluher M, Ceglarek U, Stumvoll M, Tuohy K, Diotallevi C, Vrhovsek U, Hu F, Stampfer M, Shai I. Effect of green-Mediterranean diet on intrahepatic fat: the DIRECT PLUS randomised controlled trial. Gut. 2021 Nov;70(11):2085-2095. doi: 10.1136/gutjnl-2020-323106. Epub 2021 Jan 18. PMID 33461965
- [Background] Zelicha H, Kloting N, Kaplan A, Yaskolka Meir A, Rinott E, Tsaban G, Chassidim Y, Bluher M, Ceglarek U, Isermann B, Stumvoll M, Quayson RN, von Bergen M, Engelmann B, Rolle-Kampczyk UE, Haange SB, Tuohy KM, Diotallevi C, Shelef I, Hu FB, Stampfer MJ, Shai I. The effect of high-polyphenol Mediterranean diet on visceral adiposity: the DIRECT PLUS randomized controlled trial. BMC Med. 2022 Sep 30;20(1):327. doi: 10.1186/s12916-022-02525-8. PMID 36175997
- [Background] Tsaban G, Shalev A, Katz A, Yaskolka Meir A, Rinott E, Zelicha H, Kaplan A, Wolak A, Bluher M, Stampfer MJ, Shai I. Effect of Lifestyle Modification and Green Mediterranean Diet on Proximal Aortic Stiffness. J Am Coll Cardiol. 2023 Apr 25;81(16):1659-1661. doi: 10.1016/j.jacc.2023.02.032. No abstract available. PMID 37076220
- [Background] Tsaban G, Yaskolka Meir A, Zelicha H, Rinott E, Kaplan A, Shalev A, Katz A, Brikner D, Bluher M, Ceglarek U, Stumvoll M, Stampfer MJ, Shai I. Diet-induced Fasting Ghrelin Elevation Reflects the Recovery of Insulin Sensitivity and Visceral Adiposity Regression. J Clin Endocrinol Metab. 2022 Jan 18;107(2):336-345. doi: 10.1210/clinem/dgab681. PMID 34643713
- [Background] Rinott E, Meir AY, Tsaban G, Zelicha H, Kaplan A, Knights D, Tuohy K, Scholz MU, Koren O, Stampfer MJ, Wang DD, Shai I, Youngster I. The effects of the Green-Mediterranean diet on cardiometabolic health are linked to gut microbiome modifications: a randomized controlled trial. Genome Med. 2022 Mar 10;14(1):29. doi: 10.1186/s13073-022-01015-z. PMID 35264213
- [Background] Rinott E, Youngster I, Yaskolka Meir A, Tsaban G, Zelicha H, Kaplan A, Knights D, Tuohy K, Fava F, Scholz MU, Ziv O, Rubin E, Tirosh A, Rudich A, Bluher M, Stumvoll M, Ceglarek U, Clement K, Koren O, Wang DD, Hu FB, Stampfer MJ, Shai I. Effects of Diet-Modulated Autologous Fecal Microbiota Transplantation on Weight Regain. Gastroenterology. 2021 Jan;160(1):158-173.e10. doi: 10.1053/j.gastro.2020.08.041. Epub 2020 Aug 26. PMID 32860791
- [Background] Zelicha H, Kaplan A, Yaskolka Meir A, Tsaban G, Rinott E, Shelef I, Tirosh A, Brikner D, Pupkin E, Qi L, Thiery J, Stumvoll M, Kloting N, von Bergen M, Ceglarek U, Bluher M, Stampfer MJ, Shai I. The Effect of Wolffia globosa Mankai, a Green Aquatic Plant, on Postprandial Glycemic Response: A Randomized Crossover Controlled Trial. Diabetes Care. 2019 Jul;42(7):1162-1169. doi: 10.2337/dc18-2319. Epub 2019 May 10. PMID 31076421
- [Background] Gepner Y, Golan R, Harman-Boehm I, Henkin Y, Schwarzfuchs D, Shelef I, Durst R, Kovsan J, Bolotin A, Leitersdorf E, Shpitzen S, Balag S, Shemesh E, Witkow S, Tangi-Rosental O, Chassidim Y, Liberty IF, Sarusi B, Ben-Avraham S, Helander A, Ceglarek U, Stumvoll M, Bluher M, Thiery J, Rudich A, Stampfer MJ, Shai I. Effects of Initiating Moderate Alcohol Intake on Cardiometabolic Risk in Adults With Type 2 Diabetes: A 2-Year Randomized, Controlled Trial. Ann Intern Med. 2015 Oct 20;163(8):569-79. doi: 10.7326/M14-1650. Epub 2015 Oct 13. PMID 26458258
- [Background] Dorans KS, Bazzano LA, Qi L, He H, Chen J, Appel LJ, Chen CS, Hsieh MH, Hu FB, Mills KT, Nguyen BT, O'Brien MJ, Samet JM, Uwaifo GI, He J. Effects of a Low-Carbohydrate Dietary Intervention on Hemoglobin A1c: A Randomized Clinical Trial. JAMA Netw Open. 2022 Oct 3;5(10):e2238645. doi: 10.1001/jamanetworkopen.2022.38645. PMID 36287562